CLINICAL TRIAL: NCT00311103
Title: Disability of Musculoskeletal Origin in Community-dwelling Elderly: Efficacy of a Specific Clinical Intervention.
Brief Title: Disability of Musculoskeletal Origin in Community-dwelling Elderly
Acronym: DIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spanish Foundation of Rheumatology (Other)
Collaborators: Fundacion MAPFRE (Other); Fundación Mutua Madrileña (Other); Instituto de Salud Carlos III (Other Government); La Caixa Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: PI/041582
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Musculoskeletal Diseases
Keywords: Elderly; Disability; Musculoskeletal diseases
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care in the Control Group (CG) (No Intervention): Care in the Control Group (CG): was that provided by the General Practitioners, with basic diagnostic and therapeutic procedures without specified protocols.
- Early Intervention Programa (IG) (Experimental): Early Intervention Programa (IG): Patients assigned to the intervention group after the randomization were offered an immediate appointment. Patients, who voluntarily accepted, were attended by 2 rheumatologists. The rheumatologists acted as principal care providers in regular visits, home visits and phone contacts. The visits were structured following specific proceedings for the different diagnoses based on previously demonstrated approaches. Such protocols included education and promotion of independence, pharmacological and no pharmacological treatment, and timing of diagnostic tests in a stepwise manner. The program also incorporated administrative duties such as the prescription of medication for the patients. Patients were seen as often as necessary according to the medical rheumatologist decision (until the episode of disability was medically resolved).
  Interventions: Procedure: Specific clinical care program

INTERVENTIONS:
Procedure: Specific clinical care program — The rheumatologists acted as principal care providers in regular visits, home visits and phone contacts. The visits were structured following specific proceedings for the different diagnoses based on previously demonstrated approaches. Such protocols included education and promotion of independence, pharmacological and no pharmacological treatment, and timing of diagnostic tests in a stepwise manner. The program also incorporated administrative duties such as the prescription of medication for the patients. Patients were seen as often as necessary according to the medical rheumatologist decision (until the episode of disability was medically resolved).
  Arms: Early Intervention Programa (IG)

SUMMARY:
Objectives: To assess the efficacy of an intervention program targeted to the elderly with recent-onset disability of musculoskeletal origin (DIMS), and to perform its economic evaluation.

DETAILED DESCRIPTION:
Methodology: 1) Controlled randomised intervention study (3 years). Subjects: persons older than 65 in health district 7 of Madrid with acute (< 3 months) DIMS. Intervention group patients will be attended by rheumatologists acording with clinical (diagnostic and therapeutical) protocols. Control group will receive the routine attention from the Health System. Efficacy and costs variables will be collected through monthly structured telephone interviews performed by independent personnel blinded to the intervention group. Efficacy will be measured by differences between groups regarding: 1) time to improvement in the baseline DIMS episode, 2) number of subsequent DIMS, and 3) total number of DIMS days. An economic evaluation will be performed from a societal perspective.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Musculoskeletal disorder
* Older than 64 years
* To have disability measured with a) or b):

  1. Rosser clasification: at least 4.
  2. M.Gill questionnaire: To need help from other person to dress, to tidy up itself, to walk or to stand up.
* Disability of recent onset:less than three months.(Patiens had a better functional situation before)

Exclusion Criteria:

* Recent surgery
* Dementia with no family support
* Institutionalized

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 214 (Actual)
Dates: Start 2005-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Time to improvement in the baseline recent-onset disability episode of musculoskeletal origin (DIMS) | Period of time in days until the patients recovers defined as: an improvement in at least one point in the Rosser disability level
Number of subsequent DIMS | Period of time in days until the patients recovers defined as: an improvement in at least one point in the Rosser disability level
Total number of DIMS days | Period of time in days until the patients recovers defined as: an improvement in at least one point in the Rosser disability level

SECONDARY OUTCOMES:
Direct and Indirect Costs | Period of time in days until the patients recovers defined as: an improvement in at least one point in the Rosser disability level

CONTACTS AND LOCATIONS:
Overall Officials: Juan A. Jover, MD, PhD, Principal Investigator — IMSALUD; Loreto Carmona, MD, PhD, Study Director — Spanish Foundation of Rheumatology
Locations (1):
- Hospital Clínico San Carlos, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Abasolo L, Leon L, Lajas C, Carmona L, Serra JA, Reoyo A, Rodriguez-Rodriguez L, Jover JA; APDE Group. An early intervention program for subacute physical disability related to musculoskeletal diseases in the elderly: a pilot study. Rheumatol Int. 2015 Jul;35(7):1183-91. doi: 10.1007/s00296-015-3223-3. Epub 2015 Jan 30. PMID 25634768